CLINICAL TRIAL: NCT01035749
Title: Safety and Immunogenicity Study of GSK Biologicals' Pandemic Influenza (H1N1) Candidate Vaccine (GSK2340274A) in Children Aged 10 to Less Than 18 Years
Brief Title: Study of GSK Biologicals' Pandemic Influenza (H1N1) Candidate Vaccine in Children Aged 10 to Less Than 18 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 113883
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Results first posted 2017-01-25 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2016-11

CONDITIONS: Influenza
Keywords: pandemic influenza; Clinical trial; H1N1; children
MeSH Terms: conditions — Influenza, Human | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- AREPANRIX-ADJUVANTED F1 2D GROUP (Experimental): Subjects received 2 doses of Arepanrix ™ formulation 1 adjuvanted vaccine on Day 0 and Day 182 (booster) and one dose of saline placebo on Day 21.
  Interventions: Biological: GSK Biologicals' Influenza investigational vaccine GSK2340274A; Biological: Placebo (saline)
- AREPANRIX-ADJUVANTED F2 2D GROUP (Experimental): Subjects received 2 doses of Arepanrix ™ formulation 2 adjuvanted vaccine on Day 0 and Day 182 (booster) and one dose of saline placebo on Day 21.
  Interventions: Biological: GSK Biologicals' Influenza investigational vaccine GSK2340274A; Biological: Placebo (saline)
- AREPANRIX-ADJUVANTED F2 3D GROUP (Experimental): Subjects received 3 doses of Arepanrix ™ formulation 2 adjuvanted vaccine on Day 0, Day 21 and Day 182 (booster).
  Interventions: Biological: GSK Biologicals' Influenza investigational vaccine GSK2340274A
- AREPANRIX-UNADJUVANTED F2 2D GROUP (Experimental): Subjects received 2 doses of Arepanrix ™ unadjuvanted vaccine on Day 0 and Day 182 (booster) and one dose of saline placebo on Day 21.
  Interventions: Biological: GSK Biologicals' Influenza investigational vaccine GSK2340273A; Biological: Placebo (saline)

INTERVENTIONS:
Biological: GSK Biologicals' Influenza investigational vaccine GSK2340274A — One or two doses administered intramuscularly
  Arms: AREPANRIX-ADJUVANTED F1 2D GROUP; AREPANRIX-ADJUVANTED F2 2D GROUP; AREPANRIX-ADJUVANTED F2 3D GROUP
Biological: GSK Biologicals' Influenza investigational vaccine GSK2340273A — Two doses intramuscularly
  Arms: AREPANRIX-UNADJUVANTED F2 2D GROUP
Biological: Placebo (saline) — One dose intramuscularly
  Arms: AREPANRIX-ADJUVANTED F1 2D GROUP; AREPANRIX-ADJUVANTED F2 2D GROUP; AREPANRIX-UNADJUVANTED F2 2D GROUP

SUMMARY:
The purpose of this study is to show that vaccination with a single dose of GSK Biologicals' pandemic H1N1 vaccine results in an immune response that meets or exceeds European Medicines Agency (EMEA) Committee for Medicinal Products for Human Use (CHMP) guidance criteria for a pandemic influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children 10 to < 18 years of age at the time of the first vaccination. "Less than 18 years of age" implies inclusion of adolescents who have not reached their 18th birthday as of Day 0, the day of the first vaccine dose under this protocol.
* Written informed consent obtained from the subject's parent/legally acceptable representative (LAR); written informed assent obtained from the subject if appropriate.
* Good general health as established by medical history and clinical examination before entering into the study.
* Parent/LAR access to a consistent means of telephone contact, land line or mobile, but NOT a pay phone or other multiple-user device.
* Subjects who the investigator believes that they and/or their parent(s)/LAR can and will comply with the requirements of the protocol.

Exclusion Criteria:

* Medical history of physician-confirmed infection with an A/California/7/2009 (H1N1)v-like virus.
* Previous vaccination at any time with an A/California/7/2009 (H1N1)v-like virus vaccine.
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, even if stable, are deemed by the investigator to render the potential subject or parent(s)/ LAR(s) unable/unlikely to provide accurate safety reports.
* Presence of a temperature >= 38.0ºC by any route or method, or acute symptoms greater than "mild" severity on the scheduled date of first vaccination. NOTE: The subject may be vaccinated at a later date, provided symptoms have resolved, vaccination occurs within the window specified by the protocol, and all other eligibility criteria continue to be satisfied.
* Diagnosed with cancer, or treatment for cancer, within 3 years.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Receipt of systemic glucocorticoids within 1 month prior to study enrollment (first dose of study vaccine), or any other cytotoxic or immunosuppressive drug within 6 months of study enrollment. Topical, intra-articular or inhaled glucocorticoids are allowed.
* Receipt of any immunoglobulins and/or any blood products within 6 months of study enrollment or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin are eligible if no such doses are given in the 24 hours before a study vaccination. Persons receiving prophylactic antiplatelet medications, e.g., low-dose acetylsalicylic acid, and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome within 6 weeks of receipt of seasonal influenza vaccine.
* Administration of any licensed vaccine within 30 days before the first dose of study vaccine, with the exception of seasonal influenza vaccine (which may be given within 2 weeks before the first dose of study vaccine).
* Planned administration of any A/California H1N1v-like vaccine other than the study vaccine between Day 0 and the Day 189 phlebotomy.
* Planned administration of any other vaccine not foreseen by the study protocol between Day 0 and Day 42 after the first vaccine dose, including seasonal influenza vaccine. Routine childhood vaccinations are exempted if they cannot be delayed, but they must not be administered on the same day as the H1N1 vaccine candidate.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Child in care.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 310 (Actual)
Dates: Start 2010-02-01; Primary Completion 2010-09-27 (Actual); Study Completion 2011-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- GSK Investigational Site, Tartu, Estonia
- Slovakia (8):
  - GSK Investigational Site, Cífer
  - GSK Investigational Site, Dolný Kubín
  - GSK Investigational Site, Dunajská Streda
  - GSK Investigational Site, Nová Dubnica
  - GSK Investigational Site, Nové Mesto nad Váhom
  - GSK Investigational Site, Púchov
  - GSK Investigational Site, Ružomberok
  - GSK Investigational Site, Trenčín

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 113883 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113883 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113883 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113883 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113883 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113883 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 310 subjects were enrolled in the study, all of which were vaccinated and completed the Day 42 visit.
Period: Overall Study
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Started | 66 | 66 | 68 | 110
Completed | 66 | 66 | 68 | 110
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group | Total
Number analyzed (Participants) | 66 | 66 | 68 | 110 | 310
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.6 (2.27) | 14.5 (2.2) | 14.6 (1.84) | 14.1 (2.13) | 14.19 (2.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 32 | 38 | 59 | 166
  Male | 29 | 34 | 30 | 51 | 144

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Seroconverted for HI Antibodies Against Flu A/CAL/7/09 H1N1 Strain
Description: Seroconversion defined as: - For initially seronegative subjects, antibody titre ≥ 1:40 after vaccination - For initially seropositive subjects, antibody titre after vaccination ≥ 4 fold the pre-vaccination antibody titre
Time Frame: At Day 21
Population: The analysis was performed on the ATP cohort for immunogenicity at Day21,which included all evaluated subjects for whom the injection site was known,who received the vaccine on Day0 as per protocol (PP) & for whom assay results for antibodies against A/California-like HA antigen for bloodsample taken 21days after the 1st vaccination were available.
Measure: Number; unit: Subjects
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 66 | 65 | 68 | 109
Subjects | 63 | 58 | 61 | 96

2. Primary Outcome: Number of Subjects Seroprotected for HI Antibodies Against Flu A/CAL/7/09 H1N1 Strain
Description: A seroprotected subject was defined as a subject with a serum HI titer greater than or equal to 1:40 that usually is accepted as indicating protection.
Time Frame: At Day 0 and Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 66 | 65 | 68 | 109
Subjects
  Day 0 | 28 | 35 | 30 | 49
  Day 21 | 66 | 65 | 67 | 107

3. Primary Outcome: HI Antibody Seroconversion Factors Against Flu A/CAL/7/09 H1N1 Strain
Description: Seroconversion factors were defined as the fold increase in serum HI GMTs post-vaccination compared to Day 0.
Time Frame: At Day 21
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 42,which included all evaluated subjects for whom the injection site was known, who received the vaccine/placebo on both Day 0 and 21 as PP & for whom assay results for antibodies (Abs) against A/California-like HA antigen for blood sample taken on Day 21 & 42 were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 66 | 65 | 68 | 109
Fold increase | 35.6 [26.4 to 47.9] | 18.3 [13.1 to 25.6] | 28.9 [20.4 to 41] | 25.3 [19.2 to 33.3]

4. Secondary Outcome: HI Antibody Titres Against Flu A/CAL/7/09 H1N1 Strain
Description: Antibody titres were expressed as Geometric mean titers (GMTs).
Time Frame: At Day 0 and Day 42
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 65 | 65 | 68 | 108
Titers
  Day 0 | 23.4 [16.7 to 32.9] | 33 [22.4 to 48.7] | 23.4 [16.9 to 32.4] | 22.7 [17.3 to 29.8]
  Day 42 | 646.9 [532.3 to 786.2] | 469.7 [386.9 to 570.3] | 977 [833.1 to 1145.8] | 439.6 [356 to 543]

5. Secondary Outcome: HI Antibody Titres Against Flu A/CAL/7/09 H1N1 Strain
Description: Antibody titres were expressed as GMTs.
Time Frame: At Day 0 and Day 182
Population: The analysis was performed on the ATP cohort for immunogenicity at Day182,which included all evaluated subjects for whom the injection site was known,who received the vaccine/placebo on Day0 & 21 as PP & for whom assay results for Abs against A/California-like HA antigen for bloodsample taken21,42 & 182 days after the 1st vaccination were available
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 64 | 65 | 68 | 109
Titers
  Day 0 | 22.9 [16.3 to 32] | 34.8 [23.5 to 51.5] | 23.4 [16.9 to 32.4] | 22.8 [17.4 to 29.9]
  Day 182 | 240.2 [188.1 to 306.6] | 176.1 [137.1 to 226] | 318.4 [257.8 to 393.1] | 177.2 [140.1 to 224]

6. Secondary Outcome: HI Antibody Titres Against Flu A/CAL/7/09 H1N1 Strain
Description: Antibody titres were expressed as Geometric mean titers (GMTs).
Time Frame: At Days 0, 182 and 189
Population: The analysis was performed on the ATP cohort for immunogenicity at Day189,which included all subjects for whom the injection site was known,who received the vaccine/placebo on Day0,21 & booster on Day182 as PP & for whom assay results for Abs against A/California-like HA antigen for bloodsample taken21,42,182&189D after the 1st dose were available
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 63 | 63 | 68 | 108
Titers
  Day 0 | 23.4 [16.7 to 32.9] | 33.5 [22.5 to 50.1] | 23.4 [16.9 to 32.4] | 22.5 [17.2 to 29.5]
  Day 182 | 237.7 [185.7 to 304.5] | 172.7 [133.7 to 223.2] | 318.4 [257.8 to 393.1] | 177.3 [140 to 224.7]
  Day 189 | 589.4 [506 to 686.5] | 416.7 [352.8 to 492.2] | 552.1 [474.5 to 642.5] | 273.4 [233.2 to 320.6]

7. Secondary Outcome: Number of Subjects Seroconverted for HI Antibodies Against Flu A/CAL/7/09 H1N1 Strain
Description: A seroconverted subject was defined as a subject who had either a pre-vaccination titre below 1:10 and a post-vaccination titre greater than or equal to 1:40 or a pre-vaccination titre greater than or equal to 1:10 and at least a 4-fold increase in post-vaccination titre.
Time Frame: At Day 42
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 65 | 65 | 68 | 108
Subjects | 62 | 52 | 65 | 93

8. Secondary Outcome: HI Antibody Titres Against Flu A/CAL/7/09 H1N1 Strain
Description: Antibody titers were expressed as GMTs.
Time Frame: At Day 0 and Day 21
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 66 | 65 | 68 | 109
Titers
  Day 0 | 24.1 [17.2 to 33.8] | 33 [22.4 to 48.7] | 23.4 [16.9 to 32.4] | 22.8 [17.4 to 29.9]
  Day 21 | 858.7 [714.5 to 1032] | 603.6 [493.3 to 738.5] | 676.9 [539.1 to 850] | 578.1 [466.7 to 716.1]

9. Secondary Outcome: Number of Subjects Seroconverted for HI Antibodies Against Flu A/CAL/7/09 H1N1 Strain
Description: as for outcome 7
Time Frame: At Day 182
Population: as for outcome 5
Measure: Number; unit: Subjects
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 64 | 65 | 68 | 109
Subjects | 48 | 34 | 56 | 67

10. Secondary Outcome: Number of Subjects Seroconverted for HI Antibodies Against Flu A/CAL/7/09 H1N1 Strain
Description: A seroconverted subject was defined as a subject who had either a pre-vaccination titre below 1:10 and a post-vaccination titre greater than or equal to 1:40 or a pre-vaccination titre greater than or equal to 1:10 and at least a 4-fold increase in post-vaccination titre. Day 0 was used as reference activity.
Time Frame: At Day 189
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 63 | 63 | 68 | 108
Subjects | 58 | 47 | 64 | 84

11. Secondary Outcome: Number of Subjects Seroconverted for HI Antibodies Against Flu A/CAL/7/09 H1N1 Strain
Description: A seroconverted subject was defined as a subject who had either a pre-vaccination titer below 1:10 and a post-vaccination titer greater than or equal to 1:40 or a pre-vaccination titer greater than or equal to 1:10 and at least a 4-fold increase in post-vaccination titer. Day 182 was used as reference activity.
Time Frame: At Day 189
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 63 | 63 | 68 | 108
Subjects | 17 | 18 | 9 | 11

12. Secondary Outcome: The Number of Subjects Seroprotected for HI Antibodies Against Flu A/CAL/7/09 H1N1
Description: A seroprotected subject was defined as a subject with a serum HI titre greater than or equal to 1:40 that usually is accepted as indicating protection.
Time Frame: At Day 0 and Day 42
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 65 | 65 | 68 | 108
Subjects
  Day 0 | 27 | 35 | 30 | 48
  Day 42 | 65 | 64 | 68 | 105

13. Secondary Outcome: Number of Subjects Seroprotected to HI Antibodies Against Flu A/CAL/7/09 H1N1
Description: as for outcome 12
Time Frame: At Day 0 and Day 182
Population: as for outcome 5
Measure: Number; unit: Subjects
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 64 | 65 | 68 | 109
Subjects
  Day 0 | 26 | 36 | 30 | 49
  Day 182 | 62 | 61 | 67 | 98

14. Secondary Outcome: Number of Subjects Seroprotected to HI Antibodies Against Flu A/CAL/7/09 H1N1
Description: as for outcome 2
Time Frame: At Day 0, Day 182 and Day 189
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 63 | 63 | 68 | 108
Subjects
  Day 0 | 26 | 34 | 30 | 48
  Day 182 | 61 | 59 | 67 | 97
  Day 189 | 63 | 63 | 68 | 105

15. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/CAL/7/09 H1N1
Description: GMFR (also known as the seroconversion factor, SCF) was defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the pre-vaccination reciprocal HI titer for the vaccine virus.
Time Frame: At Day 42
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 65 | 65 | 68 | 108
Fold increase | 27.6 [20.7 to 36.7] | 14.2 [10.2 to 19.8] | 41.8 [29.4 to 59.3] | 19.3 [14.7 to 25.5]

16. Secondary Outcome: GMFR for HI Antibodies Against Flu A/CAL/7/09 H1N1
Description: as for outcome 15
Time Frame: At Day 182
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 64 | 65 | 68 | 109
Fold increase | 10.5 [7.9 to 14] | 5.1 [3.7 to 6.9] | 13.6 [9.9 to 18.8] | 7.8 [5.8 to 10.3]

17. Secondary Outcome: GMFR for HI Antibodies Against Flu A/CAL/7/09 H1N1 Using Day 0 as Reference Activity
Description: as for outcome 15
Time Frame: At Day 189
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 63 | 63 | 68 | 108
Fold increase | 25.2 [17.9 to 35.3] | 12.4 [8.3 to 18.6] | 23.6 [16.6 to 33.6] | 12.1 [9.3 to 15.9]

18. Secondary Outcome: GMFR for HI Antibodies Against Flu A/CAL/7/09 H1N1 Using Day 182 as Reference Activity
Description: as for outcome 15
Time Frame: At Day 189
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 63 | 63 | 68 | 108
Fold increase | 2.5 [2 to 3.1] | 2.4 [1.9 to 3] | 1.7 [1.5 to 2] | 1.5 [1.3 to 1.8]

19. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Adverse Events (AEs)
Description: Any was defined as occurrence of any local symptom regardless of their intensity grade.Grade 3 redness and swelling was > 100 millimeter (mm) and grade 3 pain was defined as pain that prevented normal activity.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 66 | 66 | 68 | 110
Subjects
  Any pain | 52 | 48 | 61 | 51
  Grade 3 pain | 2 | 0 | 2 | 0
  Any Redness | 2 | 0 | 1 | 0
  Grade 3 Redness | 0 | 0 | 0 | 0
  Any Swelling | 4 | 1 | 6 | 1
  Grade 3 Swelling | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local AEs
Description: as for outcome 19
Time Frame: During the 7-day (Days 0-6) post-vaccination period following booster dose
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 65 | 65 | 68 | 110
Subjects
  Any Pain | 48 | 40 | 54 | 49
  Grade 3 Pain | 3 | 3 | 4 | 0
  Any Redness | 4 | 1 | 1 | 0
  Grade 3 Redness | 0 | 0 | 0 | 0
  Any Swelling | 6 | 5 | 3 | 0
  Grade 3 Swelling | 1 | 0 | 0 | 0

21. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General AEs
Description: Solicited general symptoms assessed were arthralgia, fatigue, gastrointestinal, headache, myalgia, shivering, sweating and fever (Fever = axillary temperature equal to or above 38.0 degrees Celsius (°C)). Any = any solicited general symptom reported irrespective of intensity and relationship to vaccination. Related = symptoms considered by the investigator to have a causal relationship to vaccination. Grade 3 symptoms = symptoms that prevented normal activity. Grade 3 fever = axillary temperature equal to or above (≥) 39.0°C.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 66 | 66 | 68 | 110
Subjects
  Any Arthralgia | 5 | 7 | 6 | 13
  Grade 3 Arthralgia | 0 | 0 | 0 | 0
  Related Arthralgia | 5 | 6 | 5 | 10
  Any Fatigue | 26 | 19 | 24 | 36
  Grade 3 Fatigue | 0 | 0 | 1 | 1
  Related Fatigue | 23 | 16 | 21 | 28
  Any Gastrointestinal | 5 | 3 | 9 | 8
  Grade 3 Gastrointestinal | 0 | 0 | 1 | 0
  Related Gastrointestinal | 3 | 2 | 6 | 5
  Any Headache | 27 | 21 | 39 | 45
  Grade 3 Headache | 0 | 1 | 0 | 0
  Related Headache | 23 | 16 | 27 | 31
  Any Myalgia | 17 | 20 | 28 | 21
  Grade 3 Myalgia | 0 | 0 | 0 | 0
  Related Myalgia | 16 | 17 | 23 | 16
  Any Shivering | 6 | 5 | 8 | 16
  Grade 3 Shivering | 0 | 0 | 0 | 0
  Related Shivering | 6 | 4 | 7 | 11
  Any Sweating | 6 | 8 | 11 | 15
  Grade 3 Sweating | 0 | 0 | 0 | 0
  Related Sweating | 6 | 3 | 8 | 8
  Any Fever | 2 | 0 | 1 | 3
  Grade 3 Fever | 0 | 0 | 0 | 1
  Related Fever | 2 | 0 | 1 | 2

22. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General AEs
Description: as for outcome 21
Time Frame: During the 7-day (Days 0-6) post-vaccination period following booster dose
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
  Note: 1 subject moved out of the study area thereby withdrawing from the study.
Measure: Number; unit: Subjects
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 65 | 65 | 68 | 110
Subjects
  Any Arthralgia | 13 | 8 | 12 | 8
  Grade 3 Arthralgia | 0 | 0 | 0 | 0
  Related Arthralgia | 13 | 5 | 8 | 6
  Any Fatigue | 29 | 20 | 28 | 19
  Grade 3 Fatigue | 1 | 0 | 0 | 0
  Related Fatigue | 27 | 15 | 25 | 16
  Any Gastrointestinal | 4 | 2 | 8 | 4
  Grade 3 Gastrointestinal | 1 | 0 | 0 | 0
  Related Gastrointestinal | 4 | 2 | 7 | 3
  Any Headache | 24 | 23 | 32 | 25
  Grade 3 Headache | 1 | 1 | 0 | 0
  Related Headache | 23 | 16 | 24 | 18
  Any Myalgia | 19 | 16 | 17 | 20
  Grade 3 Myalgia | 0 | 0 | 0 | 0
  Related Myalgia | 19 | 14 | 15 | 16
  Any Shivering | 9 | 13 | 15 | 9
  Grade 3 Shivering | 0 | 0 | 0 | 0
  Related Shivering | 9 | 8 | 12 | 8
  Any Sweating | 5 | 3 | 4 | 9
  Grade 3 Sweating | 0 | 0 | 0 | 0
  Related Sweating | 5 | 3 | 3 | 6
  Any Fever | 11 | 5 | 7 | 2
  Grade 3 Fever | 0 | 1 | 0 | 0
  Related Fever | 10 | 1 | 6 | 2

23. Secondary Outcome: Number of Subjects Reporting Any Medically Attended Events (MAEs)
Description: MAEs were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit or a visit to or from medical personnel (medical doctor) for any reason.
Time Frame: During the entire study period (Days 0-364) following the first vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 66 | 66 | 68 | 110
Subjects | 20 | 21 | 22 | 34

24. Secondary Outcome: Number of Subjects Reporting Potential Immune-Mediated Diseases (pIMDs)
Description: pIMDs were defined as a subset of AEs that included both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology.
Time Frame: During the entire study period (Days 0-364) following first vaccination
Population: The analysis was performed on the Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 66 | 66 | 68 | 110
Subjects | 0 | 0 | 0 | 0

25. Secondary Outcome: Number of Subjects With Normal and Abnormal Hematological and Biochemical Parameters Assessed With Respect to Normal Laboratory Ranges
Description: Subjects were categorized according to their results at pre-vaccination (PRE), Day 21, Day 42, Day 182 and Day 189 which were within normal, above normal, below the normal ranges or unknown. The laboratory parameters assessed were Alanine aminotransferase (ALAT), Aspartate aminotransferase (ASAT), Total Bilirubin, Creatinine, Hematocrit, Hemoglobin, Platelets, Blood urea nitrogen (BUN) and White blood cells (WBCs).
Time Frame: At Days 0, 21, 42, 182 and 189
Population: The analysis was performed on the Total Vaccinated cohort included all vaccinated subjects.
  Note: 1 subject moved out of the study area thereby withdrawing from the study at Days 182 and 189.
Measure: Number; unit: Subjects
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 66 | 66 | 68 | 110
Subjects
  ALAT, Day 0 Unknown | 0 | 0 | 0 | 0
  ALAT, Day 0 Below | 0 | 0 | 0 | 0
  ALAT, Day 0 Within | 65 | 65 | 66 | 108
  ALAT, Day 0 Above | 1 | 1 | 2 | 2
  ALAT, Day 21 Unknown | 0 | 0 | 0 | 0
  ALAT, Day 21 Below | 0 | 0 | 0 | 0
  ALAT, Day 21 Within | 64 | 64 | 64 | 108
  ALAT, Day 21 Above | 2 | 2 | 4 | 2
  ALAT, Day 42 Unknown | 0 | 0 | 0 | 0
  ALAT, Day 42 Below | 0 | 0 | 0 | 0
  ALAT, Day 42 Within | 64 | 66 | 66 | 104
  ALAT, Day 42 Above | 2 | 0 | 2 | 6
  ALAT, Day 182 Unknown | 0 | 0 | 0 | 0
  ALAT, Day 182 Below | 0 | 0 | 0 | 0
  ALAT, Day 182 Within | 64 | 62 | 67 | 109
  ALAT, Day 182 Above | 1 | 3 | 1 | 1
  ALAT, Day 189 Unknown | 0 | 0 | 0 | 0
  ALAT, Day 189 Below | 0 | 0 | 0 | 0
  ALAT, Day 189 Within | 64 | 61 | 67 | 110
  ALAT, Day 189 Above | 1 | 4 | 1 | 0
  ASAT, Day 0 Unknown | 0 | 0 | 0 | 0
  ASAT, Day 0 Below | 0 | 0 | 0 | 0
  ASAT, Day 0 Within | 63 | 62 | 64 | 108
  ASAT, Day 0 Above | 3 | 4 | 4 | 2
  ASAT, Day 21 Unknown | 0 | 0 | 0 | 0
  ASAT, Day 21 Below | 0 | 0 | 0 | 0
  ASAT, Day 21 Within | 61 | 61 | 63 | 104
  ASAT, Day 21 Above | 5 | 5 | 5 | 6
  ASAT, Day 42 Unknown | 0 | 0 | 0 | 0
  ASAT, Day 42 Below | 0 | 0 | 0 | 0
  ASAT, Day 42 Within | 65 | 60 | 67 | 103
  ASAT, Day 42 Above | 1 | 6 | 1 | 7
  ASAT, Day 182 Unknown | 0 | 0 | 0 | 0
  ASAT, Day 182 Below | 0 | 0 | 0 | 0
  ASAT, Day 182 Within | 63 | 61 | 67 | 110
  ASAT, Day 182 Above | 2 | 4 | 1 | 0
  ASAT, Day 189 Unknown | 0 | 0 | 0 | 0
  ASAT, Day 189 Below | 0 | 0 | 0 | 0
  ASAT, Day 189 Within | 64 | 62 | 67 | 110
  ASAT, Day 189 Above | 1 | 3 | 1 | 0
  Total Bilirubin, Day 0 Unknown | 0 | 0 | 0 | 0
  Total Bilirubin, Day 0 Below | 0 | 0 | 0 | 0
  Total Bilirubin, Day 0 Within | 21 | 22 | 19 | 36
  Total Bilirubin, Day 0 Above | 3 | 1 | 5 | 3
  Total Bilirubin, Day 21 Unknown | 0 | 0 | 0 | 0
  Total Bilirubin, Day 21 Below | 0 | 0 | 0 | 0
  Total Bilirubin, Day 21 Within | 23 | 21 | 21 | 34
  Total Bilirubin, Day 21 Above | 1 | 2 | 3 | 5
  Total Bilirubin, Day 42 Unknown | 0 | 0 | 0 | 0
  Total Bilirubin, Day 42 Below | 0 | 0 | 0 | 0
  Total Bilirubin, Day 42 Within | 22 | 21 | 20 | 37
  Total Bilirubin, Day 42 Above | 2 | 2 | 4 | 2
  Total Bilirubin, Day 182 Unknown | 0 | 0 | 0 | 0
  Total Bilirubin, Day 182 Below | 0 | 0 | 0 | 0
  Total Bilirubin, Day 182 Within | 22 | 21 | 21 | 36
  Total Bilirubin, Day 182 Above | 2 | 2 | 3 | 3
  Total Bilirubin, Day 189 Unknown | 0 | 0 | 0 | 0
  Total Bilirubin, Day 189 Below | 0 | 0 | 1 | 0
  Total Bilirubin, Day 189 Within | 22 | 22 | 21 | 35
  Total Bilirubin, Day 189 Above | 2 | 1 | 2 | 4
  Creatinine, Day 0 Unknown | 0 | 0 | 0 | 0
  Creatinine, Day 0 Below | 4 | 2 | 4 | 5
  Creatinine, Day 0 Within | 41 | 47 | 46 | 77
  Creatinine, Day 0 Above | 21 | 17 | 18 | 28
  Creatinine, Day 21 Unknown | 0 | 0 | 0 | 0
  Creatinine, Day 21 Below | 4 | 5 | 4 | 8
  Creatinine, Day 21 Within | 46 | 48 | 45 | 74
  Creatinine, Day 21 Above | 16 | 13 | 19 | 28
  Creatinine, Day 42 Unknown | 0 | 0 | 0 | 0
  Creatinine, Day 42 Below | 4 | 3 | 6 | 7
  Creatinine, Day 42 Within | 42 | 48 | 43 | 80
  Creatinine, Day 42 Above | 20 | 15 | 19 | 23
  Creatinine, Day 182 Unknown | 0 | 0 | 0 | 0
  Creatinine, Day 182 Below | 6 | 5 | 5 | 5
  Creatinine, Day 182 Within | 51 | 52 | 53 | 94
  Creatinine, Day 182 Above | 8 | 8 | 10 | 11
  Creatinine, Day 189 Unknown | 0 | 0 | 0 | 0
  Creatinine, Day 189 Below | 4 | 6 | 3 | 6
  Creatinine, Day 189 Within | 53 | 54 | 52 | 91
  Creatinine, Day 189 Above | 8 | 5 | 13 | 13
  Hematocrit, Day 0 Unknown | 0 | 0 | 0 | 0
  Hematocrit, Day 0 Below | 6 | 6 | 9 | 11
  Hematocrit, Day 0 Within | 60 | 59 | 59 | 99
  Hematocrit, Day 0 Above | 0 | 1 | 0 | 0
  Hematocrit, Day 21 Unknown | 0 | 0 | 0 | 0
  Hematocrit, Day 21 Below | 6 | 6 | 6 | 13
  Hematocrit, Day 21 Within | 59 | 60 | 61 | 95
  Hematocrit, Day 21 Above | 1 | 0 | 1 | 2
  Hematocrit, Day 42 Unknown | 0 | 0 | 0 | 0
  Hematocrit, Day 42 Below | 9 | 6 | 7 | 13
  Hematocrit, Day 42 Within | 57 | 60 | 61 | 96
  Hematocrit, Day 42 Above | 0 | 0 | 0 | 1
  Hematocrit, Day 182 Unknown | 0 | 0 | 0 | 0
  Hematocrit, Day 182 Below | 10 | 3 | 6 | 8
  Hematocrit, Day 182 Within | 55 | 61 | 62 | 102
  Hematocrit, Day 182 Above | 0 | 1 | 0 | 0
  Hematocrit, Day 189 Unknown | 0 | 0 | 0 | 0
  Hematocrit, Day 189 Below | 8 | 3 | 4 | 8
  Hematocrit, Day 189 Within | 57 | 62 | 64 | 102
  Hematocrit, Day 189 Above | 0 | 0 | 0 | 0
  Hemoglobin, Day 0 Unknown | 0 | 0 | 0 | 0
  Hemoglobin, Day 0 Below | 10 | 8 | 8 | 17
  Hemoglobin, Day 0 Within | 56 | 57 | 58 | 92
  Hemoglobin, Day 0 Above | 0 | 1 | 2 | 1
  Hemoglobin, Day 21 Unknown | 0 | 0 | 0 | 0
  Hemoglobin, Day 21 Below | 11 | 9 | 7 | 15
  Hemoglobin, Day 21 Within | 54 | 56 | 59 | 93
  Hemoglobin, Day 21 Above | 1 | 1 | 2 | 2
  Hemoglobin, Day 42 Unknown | 0 | 0 | 0 | 0
  Hemoglobin, Day 42 Below | 14 | 8 | 9 | 13
  Hemoglobin, Day 42 Within | 51 | 57 | 58 | 97
  Hemoglobin, Day 42 Above | 1 | 1 | 1 | 0
  Hemoglobin, Day 182 Unknown | 0 | 0 | 0 | 0
  Hemoglobin, Day 182 Below | 10 | 4 | 6 | 12
  Hemoglobin, Day 182 Within | 54 | 60 | 62 | 98
  Hemoglobin, Day 182 Above | 1 | 1 | 0 | 0
  Hemoglobin, Day 189 Unknown | 0 | 0 | 0 | 0
  Hemoglobin, Day 189 Below | 9 | 3 | 4 | 14
  Hemoglobin, Day 189 Within | 55 | 61 | 64 | 96
  Hemoglobin, Day 189 Above | 1 | 1 | 0 | 0
  Platelets, Day 0 Unknown | 0 | 0 | 0 | 0
  Platelets, Day 0 Below | 0 | 0 | 0 | 0
  Platelets, Day 0 Within | 24 | 23 | 24 | 39
  Platelets, Day 0 Above | 0 | 0 | 0 | 0
  Platelets, Day 21 Unknown | 0 | 0 | 0 | 0
  Platelets, Day 21 Below | 1 | 0 | 0 | 1
  Platelets, Day 21 Within | 23 | 23 | 24 | 37
  Platelets, Day 21 Above | 0 | 0 | 0 | 1
  Platelets, Day 42 Unknown | 0 | 0 | 0 | 0
  Platelets, Day 42 Below | 0 | 0 | 0 | 0
  Platelets, Day 42 Within | 24 | 23 | 24 | 39
  Platelets, Day 42 Above | 0 | 0 | 0 | 0
  Platelets, Day 182 Unknown | 0 | 0 | 0 | 0
  Platelets, Day 182 Below | 1 | 0 | 0 | 0
  Platelets, Day 182 Within | 22 | 23 | 24 | 39
  Platelets, Day 182 Above | 1 | 0 | 0 | 0
  Platelets, Day 189 Unknown | 0 | 0 | 0 | 0
  Platelets, Day 189 Below | 0 | 1 | 0 | 0
  Platelets, Day 189 Within | 23 | 22 | 24 | 39
  Platelets, Day 189 Above | 1 | 0 | 0 | 0
  BUN, Day 0 Unknown | 0 | 0 | 0 | 0
  BUN, Day 0 Below | 3 | 1 | 3 | 0
  BUN, Day 0 Within | 60 | 62 | 63 | 106
  BUN, Day 0 Above | 1 | 0 | 0 | 0
  BUN, Day 21 Unknown | 0 | 0 | 0 | 0
  BUN, Day 21 Below | 1 | 1 | 0 | 0
  BUN, Day 21 Within | 63 | 62 | 66 | 106
  BUN, Day 21 Above | 0 | 0 | 0 | 0
  BUN, Day 42 Unknown | 0 | 0 | 0 | 0
  BUN, Day 42 Below | 0 | 2 | 1 | 0
  BUN, Day 42 Within | 64 | 60 | 65 | 105
  BUN, Day 42 Above | 0 | 1 | 0 | 1
  BUN, Day 182 Unknown | 0 | 0 | 0 | 0
  BUN, Day 182 Below | 0 | 1 | 2 | 0
  BUN, Day 182 Within | 63 | 61 | 64 | 106
  BUN, Day 182 Above | 0 | 0 | 0 | 0
  BUN, Day 189 Unknown | 0 | 0 | 0 | 0
  BUN, Day 189 Below | 1 | 3 | 2 | 2
  BUN, Day 189 Within | 62 | 59 | 64 | 104
  BUN, Day 189 Above | 0 | 0 | 0 | 0
  WBCs, Day 0 Unknown | 0 | 0 | 0 | 0
  WBCs, Day 0 Below | 0 | 3 | 0 | 1
  WBCs, Day 0 Within | 64 | 54 | 62 | 104
  WBCs, Day 0 Above | 2 | 9 | 6 | 5
  WBCs, Day 21 Unknown | 0 | 0 | 0 | 0
  WBCs, Day 21 Below | 3 | 0 | 1 | 2
  WBCs, Day 21 Within | 56 | 60 | 60 | 103
  WBCs, Day 21 Above | 7 | 6 | 7 | 5
  WBCs, Day 42 Unknown | 0 | 0 | 0 | 0
  WBCs, Day 42 Below | 1 | 0 | 0 | 2
  WBCs, Day 42 Within | 63 | 64 | 64 | 103
  WBCs, Day 42 Above | 2 | 2 | 4 | 5
  WBCs, Day 182 Unknown | 0 | 0 | 0 | 0
  WBCs, Day 182 Below | 1 | 1 | 2 | 0
  WBCs, Day 182 Within | 62 | 60 | 64 | 106
  WBCs, Day 182 Above | 2 | 4 | 2 | 4
  WBCs, Day 189 Unknown | 0 | 0 | 0 | 0
  WBCs, Day 189 Below | 0 | 2 | 1 | 1
  WBCs, Day 189 Within | 62 | 60 | 61 | 105
  WBCs, Day 189 Above | 3 | 3 | 6 | 4

26. Secondary Outcome: Number of Subjects Reporting Any Unsolicited AEs
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as any symptom regardless of intensity or relationship to vaccination.
Time Frame: During the 42-day (Days 0-41) follow up period after first vaccination.
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 66 | 66 | 68 | 110
Subjects | 13 | 19 | 22 | 39

27. Secondary Outcome: Number of Subjects Reporting Any Unsolicited AEs
Description: as for outcome 26
Time Frame: During the 21-day (Days 0-20) follow-up period after booster vaccination.
Population: The analysis was performed on the Total Vaccinated cohort included all vaccinated subjects.
  Note: 1 subject moved out of the study area thereby withdrawing from the study.
Measure: Number; unit: Subjects
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 65 | 65 | 68 | 110
Subjects | 4 | 7 | 3 | 6

28. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs: medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the entire study period (Day 0 to Day 364)
Population: The analysis was performed on the Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Number analyzed (Participants) | 66 | 66 | 68 | 110
Subjects | 2 | 2 | 1 | 5

ADVERSE EVENTS:
Time Frame: SAEs were assessed throughout the study period (Days 0-364). Systematically frequent AEs were assessed 7 days after each vaccination and non-systematically frequent AEs were assessed 42 days after first vaccination and 21 days after booster vaccination.
Description: 1 subject moved out of the study area thereby withdrawing from the study in Arepanrix-adjuvanted F1 2D Group and Arepanrix-adjuvanted F2 2D Group, respectively.
Arm/Group | Arepanrix-adjuvanted F1 2D Group | Arepanrix-adjuvanted F2 2D Group | Arepanrix-adjuvanted F2 3D Group | Arepanrix-unadjuvanted F2 2D Group
Serious Adverse Events (participants affected / at risk) | 2/66 | 2/66 | 1/68 | 5/110
Other Adverse Events (participants affected / at risk) | 60/66 | 59/66 | 67/68 | 94/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arepanrix-adjuvanted F1 2D Group (N=66) | Arepanrix-adjuvanted F2 2D Group (N=66) | Arepanrix-adjuvanted F2 3D Group (N=68) | Arepanrix-unadjuvanted F2 2D Group (N=110)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Arepanrix-adjuvanted F1 2D Group (N=66) | Arepanrix-adjuvanted F2 2D Group (N=66) | Arepanrix-adjuvanted F2 3D Group (N=68) | Arepanrix-unadjuvanted F2 2D Group (N=110)
Pain (Primary phase) (General disorders) | 52 (52) | 48 (48) | 61 (61) | 51 (51) — AE reported during the primary phase of the study
Swelling (Primary phase) (General disorders) | 6 (6) | 5 (5) | 6 (6) | 1 (1) — AE reported during the Primary phase of the study
Redness (General disorders) | 4/65 (4) | 1/65 (1) | 1 (1) | 0 (0) — 1 subject moved out of the study area thereby withdrawing from the study in Flu1-F1-2D Group and Flu1-F2-2D Group, respectively.
Arthralgia (Booster phase) (General disorders) | 13/65 (13) | 8/65 (8) | 12 (12) | 8 (8) — 1 subject moved out of the study area thereby withdrawing from the study in Flu1-F1-2D Group and Flu1-F2-2D Group, respectively. AE reported during the Booster phase of the study.
Fatigue (Booster phase) (General disorders) | 29/65 (29) | 20/65 (20) | 28 (28) | 36 (36) — 1 subject moved out of the study area thereby withdrawing from the study in Flu1-F1-2D Group and Flu1-F2-2D Group, respectively. AE reported during the Booster phase of the study.
Headache (Primary phase) (General disorders) | 27 (27) | 21 (21) | 39 (39) | 45 (45) — AE reported during the Primary phase of the study.
Myalgia (Booster phase) (General disorders) | 19/65 (19) | 16/65 (16) | 17 (17) | 20 (20) — 1 subject moved out of the study area thereby withdrawing from the study in Flu1-F1-2D Group and Flu1-F2-2D Group, respectively. AE reported during the Booster phase of the study.
Shivering (Primary phase) (General disorders) | 6 (6) | 5 (5) | 8 (8) | 16 (16) — AE reported during the Primary phase of the study.
Sweating (Primary phase) (General disorders) | 6 (6) | 8 (8) | 11 (11) | 15 (15) — AE was reported during the Primary phase of the study.
Pain (Booster phase) (General disorders) | 48/65 (48) | 40/65 (40) | 54 (54) | 49 (49) — 1 subject moved out of the study area thereby withdrawing from the study in Flu1-F1-2D Group and Flu1-F2-2D Group, respectively. AE reported during the Booster phase of the study
Swelling (Booster phase) (General disorders) | 6/65 (6) | 5/65 (5) | 3 (3) | 0 (0) — 1 subject moved out of the study area thereby withdrawing from the study in Flu1-F1-2D Group and Flu1-F2-2D Group, respectively. AE reported during the Booster phase of the study.
Arthralgia (Primary phase) (General disorders) | 5 (5) | 7 (7) | 6 (6) | 13 (13) — AE reported during the Primary phase of the study.
Fatigue (Primary phase) (General disorders) | 26 (26) | 19 (19) | 24 (24) | 36 (36) — AE was reported during the Primary phase of the study.
Headache (Booster phase) (General disorders) | 24/65 (24) | 23/65 (23) | 32 (32) | 25 (25) — 1 subject moved out of the study area thereby withdrawing from the study in Flu1-F1-2D Group and Flu1-F2-2D Group, respectively. AE reported during the Booster phase of the study.
Myalgia (Primary phase) (General disorders) | 17 (17) | 20 (20) | 28 (28) | 21 (21) — AE reported during the Primary phase of the study.
Shivering (Booster phase) (General disorders) | 9/65 (9) | 13/65 (13) | 15 (15) | 9 (9) — 1 subject moved out of the study area thereby withdrawing from the study in Flu1-F1-2D Group and Flu1-F2-2D Group, respectively. AE reported during the Booster phase of the study.
Sweating (Booster phase) (General disorders) | 5/65 (5) | 3/65 (3) | 4 (4) | 9 (9) — 1 subject moved out of the study area thereby withdrawing from the study in Flu1-F1-2D Group and Flu1-F2-2D Group, respectively. AE was reported during the Booster phase of the study.
Gastrointestinal (Primary phase) (Gastrointestinal disorders) | 5 (5) | 3 (3) | 9 (9) | 8 (8) — AE reported during the Primary phase of the study.
Gastrointestinal (Booster phase) (Gastrointestinal disorders) | 4/65 (4) | 2/65 (2) | 8 (8) | 5 (5) — 1 subject moved out of the study area thereby withdrawing from the study in Flu1-F1-2D Group and Flu1-F2-2D Group, respectively. AE was reported during the Booster phase of the study.
Fever (Infections and infestations) | 11/65 (11) | 5/65 (5) | 7 (7) | 2 (2) — 1 subject moved out of the study area thereby withdrawing from the study in Flu1-F1-2D Group and Flu1-F2-2D Group, respectively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.